CLINICAL TRIAL: NCT04674904
Title: Effects of Dry Needling on Pain, Range of Motion and Function in Patient With Upper Cross Syndrome
Brief Title: Effects of Dry Needling in Patients With Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/LHR/20/1049 Komal Arooj
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Neck Syndrome
Keywords: Dry needling, upper cross syndrome, VAS, NDI, goniometry
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Dry Needling
  Interventions: Other: Dry Needling
- Group B (Active Comparator): Hot pack , TENS , Stretching
  Interventions: Other: Hot pack , TENS , Stretching

INTERVENTIONS:
Other: Dry Needling — Dry needling on Upper trapezius, Levator Scapulae, Sternocledomastoid , Pectorals major and minor and rhomboids for 10 min
  Arms: Group A
Other: Hot pack , TENS , Stretching — Treatments are
  1. Hot Pack for 15 minutes
  2. TENS for 10 minutes
  3. Stretching
  The third treatment which is Stretching will be given one time on each muscle (tight upper trap, Levator Scapulae, Sternocledomastoid , Pectorals major and minor and rhomboids) of upper spine
  Arms: Group B

SUMMARY:
The study will be done to evaluate the effectiveness of dry needling of muscles involved in Upper Cross Syndrome. Muscles involved in upper cross syndrome are tight upper trap, Levator Scapulae, Sternocledomastoid , Pectorals major and minor and rhomboids. Physical assessment of trigger points will locate the target area for dry needling. After pre treatment measurements, dry needling will be performed to treatment group and stretching, hot pack and tens will be apply in control group. Study design will be randomized controlled trial and sample size will be 34 participants. Data will be collected from Riphah Rehabilitation Center. Patients of 20-50 years old with UCS diagnosed through observation and physical examination will be included. Patients with systemic soft tissue and bony diseases will be excluded. Intervention duration will be two session of DNT with two weeks routine management. Basic tools will be Visual analog scale (VAS), Neck Disability Index (NDI) and Goniometry

DETAILED DESCRIPTION:
Dry needling is relatively new method for the management of musculoskeletal pain.Different methods of dry needling, its effectiveness, and physiologic and adverse effects are discussed. Dry needling is a treatment modality that is minimally invasive, cheap, easy to learn with appropriate training, and carries a low risk. The deep method of dry needling has been shown to be more effective than the superficial one for the treatment of pain associated with myofascial trigger points. However, over areas with potential risk of significant adverse events, such as lungs and large blood vessels, we suggest using the superficial technique, which has also been shown to be effective. Questionnaire for assessing the improvement in quality of life is by NDI and ranges like neck flexion/extension, side bending and rotation will be measured by standard goniometry. Neck disability index will use to check the patient's ability to perform his ADL before and after the treatment/control. Data will be collected from Riphah rehab center. Assessed patients of UCS of age 20 to 50 will be the targeted population of this study. Patients with systematic and bony disease excluded from the study. Population having stiff upper back, tight trap and stiff upper thoracic spine have UCS. Ethical guidelines will be followed for both treatment and control group. SPSS version 21 will be use for data analysis with sample size of 34 participants, 17 participants each group that will randomly allocated in treatment/control group.

ELIGIBILITY:
Inclusion Criteria:

* Stiffness and gradual pain in neck and shoulder
* Pain due to Postural Dysfunction
* Trauma or insidious onset

Exclusion Criteria:

* Any systemic soft tissue and bony disease.
* Patient with spinal tuberculosis, spinal fractures, pregnancy, cancer.
* Any recent surgery.
* Patient with any cervical or thoracic problem.
* Patients with any other serious pathology/red flags

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 2nd Week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured

SECONDARY OUTCOMES:
Neck Disability Index Questionnaire | 2nd Week
  Neck disability index is a self report questionnaire use to determine how neck pain effects the patients daily life and to assess the self rated disability of patients with neck pain. Area of assessment are activities of daily life, attention ,work memory ,functional mobility ,pain ,occupational performance ,quality of life and sleep. Totally based on patient reported outcome

OTHER OUTCOMES:
Goniometer | 2nd Week
  Goniometer is an instrument particularly useful when measuring the spine where you can use it to measure flexion, extension, side bending and rotation quickly and easily

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Sheikh Zaid Hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Gerber LH, Shah J, Rosenberger W, Armstrong K, Turo D, Otto P, Heimur J, Thaker N, Sikdar S. Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects With Chronic Myofascial Pain. PM R. 2015 Jul;7(7):711-718. doi: 10.1016/j.pmrj.2015.01.020. Epub 2015 Feb 4. PMID 25661462
- [Background] Kalichman L, Vulfsons S. Dry needling in the management of musculoskeletal pain. J Am Board Fam Med. 2010 Sep-Oct;23(5):640-6. doi: 10.3122/jabfm.2010.05.090296. PMID 20823359
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Gonzalez-Perez LM, Infante-Cossio P, Granados-Nunez M, Urresti-Lopez FJ. Treatment of temporomandibular myofascial pain with deep dry needling. Med Oral Patol Oral Cir Bucal. 2012 Sep 1;17(5):e781-5. doi: 10.4317/medoral.17822. PMID 22549679
- [Background] Ahmad Z, ur Rehman S, Ahmad S, Afzal MF. Effects of combined manual postural correction technique in patient with upper cross syndrome. Rawal Medical Journal. 2019;44(3):486-9.
- [Background] Thacker D, Jameson J, Baker J, Divine J, Unfried A. Management of upper cross syndrome through the use of active release technique and prescribed exercises. Logan College of Chiropractic. 2011 Apr
- [Background] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789